CLINICAL TRIAL: NCT07329244
Title: Clinical Evaluation of Graphene-Reinforced CAD/CAM Indirect Restorations in Molars Affected by Molar-Incisor Hypomineralization (MIH) in Adolescents: A Clinical Study
Brief Title: Graphene-Reinforced CAD/CAM Restorations for MIH-Affected Molars in Adolescents: A Prospective Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Clínica Odontologica de la Universidad de Barcelona ( UB) (Unknown)
Responsible Party: Principal Investigator, Luis Carlos Garza Garza, Restorative and Prosthodontics MSc., Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 64/2025
Record Dates: First submitted 2025-11-30; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Tooth Demineralization; Tooth Sensitivity; Enamel Mineralization Disorders; Tooth Sensitivity After Composite Restorations; Tooth Eruption Disorder; Indirect Restoration
Keywords: molar-incisor hypomineralization; MIH; enamel defects; indirect restorations; minimally invasive dentistry; adhesive dentistry
MeSH Terms: conditions — Tooth Demineralization; Dentin Sensitivity; Molar Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Graphene-Reinforced CAD/CAM Indirect Restoration (Experimental): Minimally invasive preparation, composite base build-up when indicated, adhesive protocol with total-etch technique, CAD/CAM fabrication using graphene-reinforced polymer (G-CAM®), adhesive cementation under rubber dam isolation, finishing and polishing, and follow-up at 1 week, 3, 6, and 12 months.
  Interventions: Device: Graphene-reinforced CAD/CAM polymer (G-CAM®)

INTERVENTIONS:
Device: Graphene-reinforced CAD/CAM polymer (G-CAM®) — Graphene-reinforced CAD/CAM polymer (G-CAM®) used for the fabrication of indirect inlay, onlay, or overlay restorations in permanent molars affected by molar-incisor hypomineralization (MIH). Restorations are fabricated using a digital CAD/CAM workflow and adhesively cemented under rubber dam isolation according to the study protocol.

SUMMARY:
This study evaluates the clinical performance, marginal integrity, surface wear, color stability, and postoperative sensitivity of graphene-reinforced CAD/CAM indirect restorations (inlays, onlays, overlays) in molars affected by moderate to severe Molar-Incisor Hypomineralization (MIH) in adolescents. A total of 30 patients aged 10-16 years will receive minimally invasive indirect restorations fabricated from a nano-reinforced graphene polymer (G-CAM®). Clinical outcomes will be assessed using FDI criteria, VAS sensitivity scores, patient satisfaction, and digital 3D scans over a 12-month follow-up. The study aims to determine clinical acceptability and safety compared with historical outcomes reported for composite and lithium-disilicate indirect restorations.

DETAILED DESCRIPTION:
This is a prospective, single-arm, monocentric clinical trial designed to assess the functional performance, marginal adaptation, wear behavior, postoperative sensitivity, and structural preservation of graphene-reinforced CAD/CAM restorations placed on MIH-affected molars in adolescents aged 10-16 years. MIH lesions present compromised enamel quality with increased porosity, susceptibility to post-eruptive breakdown, and frequent hypersensitivity, making conventional restorative approaches less predictable.

Minimally invasive preparations will be performed followed by adhesive placement of graphene-reinforced CAD/CAM indirect restorations fabricated through a fully digital workflow (intraoral scanning, CAD design, CAM milling). Evaluations will be performed at baseline, 48 h, 1, 3, 6, and 12 months. Primary variables include global and domain-specific FDI clinical scores (marginal integrity, surface roughness, color stability, fractures/chipping, proximal contact, occlusion/function, soft tissue response) and postoperative sensitivity measured using a Visual Analog Scale (VAS). Secondary outcomes include patient satisfaction, tooth vitality, digital volumetric analysis of structural preservation, survival of restorations, and efficiency of the digital workflow.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10-16 years.
* Permanent molars with moderate or severe MIH (EAPD criteria).
* Vital and restorable teeth.
* Ability to attend follow-up visits.
* Informed consent from guardian + assent from the minor.

Exclusion Criteria:

* Fluorosis, amelogenesis imperfecta, or other enamel defects.
* Severe bruxism not controlled.
* Active extensive caries or irreversible pulpitis.
* Systemic conditions affecting enamel or healing.
* Hypersensitivity/allergy to materials/adhesives.
* Use of analgesics/AINEs <24 h before baseline VAS.

  * Orthodontic bands on the study molar.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-04-23 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Acceptability Assessed by the FDI World Dental Federation Clinical Criteria Score | 12 months after restoration placement
  Clinical performance of the indirect CAD/CAM graphene-reinforced restoration will be evaluated using the FDI World Dental Federation Clinical Criteria.
  Each domain is scored on a 1-5 ordinal scale, where:
  1. = Clinically excellent (best outcome)
  2. = Clinically good
  3. = Clinically acceptable
  4. = Clinically unsatisfactory
  5. = Clinically poor (worst outcome)
  Domains assessed:
  Marginal integrity
  Surface roughness/wear
  Color stability
  Fractures/chipping
  Proximal contact
  Occlusion/function
  Soft tissue response
  Higher scores indicate worse clinical performance. Data will be reported as mean score per domain and global acceptability.
Postoperative Sensitivity Measured by Visual Analog Scale (VAS 0-10) | Baseline (preoperative), 48 hours, 1 month, 3 months, 6 months, and 12 months
  Postoperative sensitivity to cold and mastication will be measured on a 0-10 Visual Analog Scale (VAS), where:
  0 = No pain (best outcome)
  10 = Worst imaginable pain (worst outcome)
  Higher scores indicate worse sensitivity.

SECONDARY OUTCOMES:
Patient Satisfaction Measured by 5-Point Likert Scale | 1 month, 3 months, 6 months, and 12 months
  Patient satisfaction with the restoration will be measured on a Likert scale from 1 to 5, where:
  1. = Very dissatisfied (worst outcome)
  2. = Dissatisfied
  3. = Neutral
  4. = Satisfied
  5. = Very satisfied (best outcome)
  Higher scores indicate higher satisfaction.
Change in Tooth Structure Volume Measured by 3D Intraoral Scan Superimposition (mm³) | Baseline and 12 months
  Structural preservation will be evaluated by comparing preoperative and 12-month postoperative 3D intraoral scans.
  The primary metric is change in tooth volume (mm³) obtained through digital superimposition.
  Decreased volume indicates structural loss; minimal change indicates better preservation.
  Lower volume loss indicates better structural preservation.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Esthetic BCN, Sarrià-Sant Gervasi, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers. The study involves pediatric participants, and all data will be pseudonymized and stored in secure, access-restricted servers according to GDPR and local ethics requirements. Because the dataset is small, contains sensitive clinical information from minors, and is collected within a single clinical center, sharing IPD may increase the risk of re-identification. Therefore, IPD will not be made available outside the research team.

REFERENCES:
- [Background] Mendonca FL, Grizzo IC, Alencar CRB, Rios D. Restorative Therapy of MIH-Affected Molars. Monogr Oral Sci. 2024;32:236-260. doi: 10.1159/000538890. Epub 2024 Jul 1. PMID 39321762
- [Background] Somani C, Taylor GD, Garot E, Rouas P, Lygidakis NA, Wong FSL. An update of treatment modalities in children and adolescents with teeth affected by molar incisor hypomineralisation (MIH): a systematic review. Eur Arch Paediatr Dent. 2022 Feb;23(1):39-64. doi: 10.1007/s40368-021-00635-0. Epub 2021 Jun 10. PMID 34110615

DOCUMENTS (2):
  • Study Protocol (2025-12-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT07329244/Prot_000.pdf
  • Informed Consent Form (2025-12-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT07329244/ICF_001.pdf